CLINICAL TRIAL: NCT07101172
Title: A Simple Approach to Managing Anxiety and Pain During Prostate Biopsy: Effectiveness of Stress Ball Application
Brief Title: The Effectiveness of Stress Ball in Managing Anxiety and Pain During Prostate Biopsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Zehra UNAL, assistant professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HititZU
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Pain; Prostate Biopsy
Keywords: Anxiety; Pain; Prostate Biopsy; Stress Ball
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball (Experimental)
  Interventions: Procedure: stress ball
- control group (No Intervention)

INTERVENTIONS:
Procedure: stress ball — Patients will be provided with an explanation, and verbal and written consent will be obtained. A patient identification form will be completed 10 minutes before the procedure. Pain levels will be determined with a pre-test VAS, anxiety levels will be determined with a STAI-S, and vital signs will be measured and recorded. The patient will be undressed and helped into a surgical gown to protect their privacy. The patient will be placed in a left lateral position on a stretcher with both legs drawn up toward their abdomen. The environment will be quiet and free from external stimuli. During the biopsy procedure, the patient will be asked to squeeze and release the Stre ball once every five counts for 10 minutes. Because blood pressure may drop or dizziness may occur after the procedure, the patient will be taken to the recovery room and monitored for bleeding. Fifteen minutes after the procedure, the severity of pain and anxiety levels during the procedure will be determined, and vital
  Arms: Stress Ball

SUMMARY:
This study aimed to determine the effectiveness of stress ball application in the management of anxiety and pain during prostate biopsy.

DETAILED DESCRIPTION:
The aim of this study was to determine the effectiveness of stress ball application in managing anxiety and pain during prostate biopsy.

This experimental study was performed with experimental-control group (N=66) patients.Data will be collected using the "Personal Information Form", "Visual Analog Scale (VAS)", "State Anxiety Inventory (STAI-S)" and "Patient Follow-up Form".

ELIGIBILITY:
Inclusion Criteria:

* Patients who come to the Urology Service for a prostate biopsy, are willing to participate in the study, are over 18 years of age, are conscious, literate, have no visual or hearing impairments, no psychiatric diagnoses or neurological problems, are undergoing a prostate biopsy for the first time, and do not have weakness in their hands or arms to squeeze a ball will be included.

Exclusion Criteria:

* Patients who do not volunteer to participate in the study, who wish to withdraw from the study, who are under 18 years of age, who are unconscious, illiterate, visually or hearing impaired, who have a psychiatric diagnosis or neurological problem, who have previously had a prostate biopsy, and who have weakness in the hand or arm for the ability to squeeze a ball will be excluded from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 12 months
  Personal Information Form : This form, developed by the researcher based on literature, includes the age, education level, marital status, employment status, income level, daily pain coping strategies, stress coping strategies, previous surgery history, and whether patients are aware of prostate biopsy. It consists of nine questions . It will be used to determine the individual characteristics of the patient.
Visual Analog Scale (VAS) | 12 months
  Visual Analog Scale (VAS) : This scale is used to assess the severity of pain. It is usually a 10 cm long horizontal or vertical line that begins with "No pain" and ends with "Unbearable pain." It will be used to determine the patient's pain intensity.
State Anxiety Inventory (STAI-S) | 12 months
  State Anxiety Inventory (STAI-S) (Appendix 3): The State Anxiety Inventory has two subscales, each consisting of 20 items. The State Anxiety Inventory (STAI-S) describes how individuals feel under different circumstances and in the moment, while the Trait Anxiety Inventory (STAI-T) describes how they generally feel in their lives. The inventory is a 4-point Likert-type scale, with ratings based on the severity of the emotions and behaviors in the State and Trait Anxiety Subscales. According to the results, average anxiety scores range from 36 to 41, with scores above indicating high anxiety and below indicating low anxiety. It will be used to determine the patient's anxiety level.
Patient Follow-up Form | 12 months
  Patient Follow-up Form: This is the form created to record the vital signs of the patients [pulse, respiratory rate, systolic blood pressure (SBP), diastolic blood pressure (DBP) and oxygen saturation values (SpO2)) measured by the researcher before and after the procedure. It will be used to monitor and evaluate the patient's vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR